CLINICAL TRIAL: NCT06848153
Title: Effect of Plantar Vibration on Ankle Proprioception in Stroke Patients
Brief Title: Effect of Plantar Vibration in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Omer Dursun, Asst. Prof., Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BEUFTR-7
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Proprioception
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The evaluator and the researcher administering the plantar vibration intervention will be different. Patients will be blinded to their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Vibration Group (Placebo Comparator): In addition to the conventional treatment program, the placebo plantar vibration application will be applied to the plantar region of the patients in the placebo group. For the application, the local vibration device will be moved without touching the patient's skin while it is operational. The placebo plantar vibration will be applied for 30 minutes each day over 3 consecutive days.
  Interventions: Other: Placebo Plantar Vibration
- Local Vibration Intervention Group (Experimental): In addition to the conventional treatment program, the patients in this group will receive plantar vibration application on the affected plantar region, utilizing a frequency of 100 Hz. The plantar vibration will be applied for 30 minutes each day over 3 consecutive days.
  Interventions: Other: Plantar Vibration

INTERVENTIONS:
Other: Plantar Vibration — The patients in the study group will receive plantar vibration intervention with a frequency of 100 Hz on the affected plantar region for 30 minutes each day over 3 consecutive days.
  Arms: Local Vibration Intervention Group
Other: Placebo Plantar Vibration — The patients in the placebo group will receive placebo plantar vibration intervention with a frequency of 100 Hz on the affected plantar region, without touching the skin, for 30 minutes each day over 3 consecutive days.
  Arms: Placebo Vibration Group

SUMMARY:
The aim of the study is to investigate the effect of plantar vibration on the ankle proprioception of patients with stroke.

DETAILED DESCRIPTION:
The study, utilizing a randomized placebo controlled design, is planned to be conducted on a minimum of 34 patients with stroke who meet the inclusion and exclusion criteria. Patients included in the study will be randomly assigned to receive plantar vibration or placebo plantar vibration interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Two months or longer elapsed since the stroke,
2. A Mini-Mental State Examination score of 24 or higher,
3. Being between 45 and 75 years of age,
4. Having a Brunnstrom stage of 4 or above,
5. Ability to stand independently for 20 seconds or more,
6. Ability to walk independently for 10 meters, using assistive devices or orthoses if necessary.

Exclusion Criteria:

1. The presence of severe osteoarthritis in the lower extremity,
2. The presence of cancer or diabetic neuropathy,
3. The presence of vestibular disorder,
4. The presence of lower extremity ulceration or amputation,
5. Hemodynamic instability,
6. The presence of other neurological disorders (such as multiple sclerosis, Parkinson's disease),
7. Having experienced an acute lower extremity injury in the last six weeks,
8. History of lower extremity surgery,
9. Alcohol consumption in the last 24 hours
10. Posterior circulation stroke involving the basilar artery or cerebellum

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Ankle Proprioception | Change from baseline ankle proprioception immediately and one week after the intervention
  The effect of plantar vibration on ankle proprioception will be evaluated using the Cybex isokinetic dynamometer. The device will analyze the passive joint position sense of the ankle in various positions.

CONTACTS AND LOCATIONS:
Overall Officials: ömer dursun, Asst. Prof., Principal Investigator — Bitlis Eren University; burak mavuş, M.Sc., Principal Investigator — Bolu Abant İzzet Baysal Physiotherapy and Rehabilitation Training and Research Hospital
Locations (1):
- Bolu İzzet Baysal Fizik Tedavi ve Rehabilitasyon Eğitim ve Araştırma Hastanesi, Bolu, Merkez, Turkey (Türkiye)

REFERENCES:
- [Background] del Pozo-Cruz B, Adsuar JC, Parraca JA, del Pozo-Cruz J, Olivares PR, Gusi N. Using whole-body vibration training in patients affected with common neurological diseases: a systematic literature review. J Altern Complement Med. 2012 Jan;18(1):29-41. doi: 10.1089/acm.2010.0691. Epub 2012 Jan 10. PMID 22233167
- [Background] Speelman AD, van de Warrenburg BP, van Nimwegen M, Petzinger GM, Munneke M, Bloem BR. How might physical activity benefit patients with Parkinson disease? Nat Rev Neurol. 2011 Jul 12;7(9):528-34. doi: 10.1038/nrneurol.2011.107. PMID 21750523
- [Background] Wenning GK, Ebersbach G, Verny M, Chaudhuri KR, Jellinger K, McKee A, Poewe W, Litvan I. Progression of falls in postmortem-confirmed parkinsonian disorders. Mov Disord. 1999 Nov;14(6):947-50. doi: 10.1002/1531-8257(199911)14:63.0.co;2-o. PMID 10584668
- [Background] Arene N, Hidler J. Understanding motor impairment in the paretic lower limb after a stroke: a review of the literature. Top Stroke Rehabil. 2009 Sep-Oct;16(5):346-56. doi: 10.1310/tsr1605-346. PMID 19903653
- [Background] Lamb SE, Ferrucci L, Volapto S, Fried LP, Guralnik JM; Women's Health and Aging Study. Risk factors for falling in home-dwelling older women with stroke: the Women's Health and Aging Study. Stroke. 2003 Feb;34(2):494-501. PMID 12574566
- [Background] Tyson SF, Hanley M, Chillala J, Selley A, Tallis RC. Balance disability after stroke. Phys Ther. 2006 Jan;86(1):30-8. doi: 10.1093/ptj/86.1.30. PMID 16386060
- [Background] Yates JS, Lai SM, Duncan PW, Studenski S. Falls in community-dwelling stroke survivors: an accumulated impairments model. J Rehabil Res Dev. 2002 May-Jun;39(3):385-94. PMID 12173758
- [Background] Khalifeloo M, Naghdi S, Ansari NN, Akbari M, Jalaie S, Jannat D, Hasson S. A study on the immediate effects of plantar vibration on balance dysfunction in patients with stroke. J Exerc Rehabil. 2018 Apr 26;14(2):259-266. doi: 10.12965/jer.1836044.022. eCollection 2018 Apr. PMID 29740561
- [Background] Chen JC, Shaw FZ. Progress in sensorimotor rehabilitative physical therapy programs for stroke patients. World J Clin Cases. 2014 Aug 16;2(8):316-26. doi: 10.12998/wjcc.v2.i8.316. PMID 25133141
- [Background] Pollock A, Baer G, Campbell P, Choo PL, Forster A, Morris J, Pomeroy VM, Langhorne P. Physical rehabilitation approaches for the recovery of function and mobility following stroke. Cochrane Database Syst Rev. 2014 Apr 22;2014(4):CD001920. doi: 10.1002/14651858.CD001920.pub3. PMID 24756870
- [Background] Geurts AC, de Haart M, van Nes IJ, Duysens J. A review of standing balance recovery from stroke. Gait Posture. 2005 Nov;22(3):267-81. doi: 10.1016/j.gaitpost.2004.10.002. Epub 2004 Dec 7. PMID 16214666
- [Background] Sajedifar M, Fakhari Z, Naghdi S, Nakhostin Ansari N, Honarpisheh R, Nakhostin-Ansari A. Comparison of the immediate effects of plantar vibration of both feet with the plantar vibration of the affected foot on balance in patients with stroke: Preliminary findings. J Bodyw Mov Ther. 2023 Oct;36:45-49. doi: 10.1016/j.jbmt.2023.06.001. Epub 2023 Jun 5. PMID 37949597
- [Background] Onal B, Sertel M, Karaca G. Effect of plantar vibration on static and dynamic balance in stroke patients: a randomised controlled study. Physiotherapy. 2022 Sep;116:1-8. doi: 10.1016/j.physio.2022.02.002. Epub 2022 Feb 14. PMID 35462214
- [Background] Onal B, Karaca G, Sertel M. Immediate Effects of Plantar Vibration on Fall Risk and Postural Stability in Stroke Patients: A Randomized Controlled Trial. J Stroke Cerebrovasc Dis. 2020 Dec;29(12):105324. doi: 10.1016/j.jstrokecerebrovasdis.2020.105324. Epub 2020 Sep 28. PMID 32992184
- [Background] Lee SW, Cho KH, Lee WH. Effect of a local vibration stimulus training programme on postural sway and gait in chronic stroke patients: a randomized controlled trial. Clin Rehabil. 2013 Oct;27(10):921-31. doi: 10.1177/0269215513485100. Epub 2013 Jul 1. PMID 23818408
- [Background] Picelli A, Tamburin S, Cavazza S, Scampoli C, Manca M, Cosma M, Berto G, Vallies G, Roncari L, Melotti C, Santilli V, Smania N. Relationship between ultrasonographic, electromyographic, and clinical parameters in adult stroke patients with spastic equinus: an observational study. Arch Phys Med Rehabil. 2014 Aug;95(8):1564-70. doi: 10.1016/j.apmr.2014.04.011. Epub 2014 May 2. PMID 24792138
- [Background] Cho KH, Lee HJ, Lee WH. Intra- and inter-rater reliabilities of measurement of ultrasound imaging for muscle thickness and pennation angle of tibialis anterior muscle in stroke patients. Top Stroke Rehabil. 2017 Jul;24(5):368-373. doi: 10.1080/10749357.2017.1285745. Epub 2017 Feb 15. PMID 28198659
- [Background] Picelli A, Bonetti P, Fontana C, Barausse M, Dambruoso F, Gajofatto F, Girardi P, Manca M, Gimigliano R, Smania N. Is spastic muscle echo intensity related to the response to botulinum toxin type A in patients with stroke? A cohort study. Arch Phys Med Rehabil. 2012 Jul;93(7):1253-8. doi: 10.1016/j.apmr.2012.02.005. Epub 2012 Apr 12. PMID 22502807
- [Background] Heckmatt JZ, Leeman S, Dubowitz V. Ultrasound imaging in the diagnosis of muscle disease. J Pediatr. 1982 Nov;101(5):656-60. doi: 10.1016/s0022-3476(82)80286-2. PMID 7131136
- [Background] Pillen S, van Keimpema M, Nievelstein RA, Verrips A, van Kruijsbergen-Raijmann W, Zwarts MJ. Skeletal muscle ultrasonography: Visual versus quantitative evaluation. Ultrasound Med Biol. 2006 Sep;32(9):1315-21. doi: 10.1016/j.ultrasmedbio.2006.05.028. PMID 16965971
- [Background] Picelli A, Bonetti P, Fontana C, Barausse M, Dambruoso F, Gajofatto F, Tamburin S, Girardi P, Gimigliano R, Smania N. Accuracy of botulinum toxin type A injection into the gastrocnemius muscle of adults with spastic equinus: manual needle placement and electrical stimulation guidance compared using ultrasonography. J Rehabil Med. 2012 May;44(5):450-2. doi: 10.2340/16501977-0970. PMID 22549655
- [Background] Gao F, Grant TH, Roth EJ, Zhang LQ. Changes in passive mechanical properties of the gastrocnemius muscle at the muscle fascicle and joint levels in stroke survivors. Arch Phys Med Rehabil. 2009 May;90(5):819-26. doi: 10.1016/j.apmr.2008.11.004. PMID 19406302
- [Background] Maganaris CN, Baltzopoulos V. Predictability of in vivo changes in pennation angle of human tibialis anterior muscle from rest to maximum isometric dorsiflexion. Eur J Appl Physiol Occup Physiol. 1999 Feb;79(3):294-7. doi: 10.1007/s004210050510. PMID 10048637
- [Background] Manal K, Roberts DP, Buchanan TS. Optimal pennation angle of the primary ankle plantar and dorsiflexors: variations with sex, contraction intensity, and limb. J Appl Biomech. 2006 Nov;22(4):255-63. doi: 10.1123/jab.22.4.255. PMID 17293622
- [Background] Raj IS, Bird SR, Shield AJ. Reliability of ultrasonographic measurement of the architecture of the vastus lateralis and gastrocnemius medialis muscles in older adults. Clin Physiol Funct Imaging. 2012 Jan;32(1):65-70. doi: 10.1111/j.1475-097X.2011.01056.x. Epub 2011 Sep 25. PMID 22152081
- [Background] Filippi GM, Rodio A, Fattorini L, Faralli M, Ricci G, Pettorossi VE. Plastic changes induced by muscle focal vibration: A possible mechanism for long-term motor improvements. Front Neurosci. 2023 Feb 22;17:1112232. doi: 10.3389/fnins.2023.1112232. eCollection 2023. PMID 36908788
- [Background] Good DC, Bettermann K, Reichwein RK. Stroke rehabilitation. Continuum (Minneap Minn). 2011 Jun;17(3 Neurorehabilitation):545-67. doi: 10.1212/01.CON.0000399072.61943.38. PMID 22810867
- [Background] Filippi GM, Brunetti O, Botti FM, Panichi R, Roscini M, Camerota F, Cesari M, Pettorossi VE. Improvement of stance control and muscle performance induced by focal muscle vibration in young-elderly women: a randomized controlled trial. Arch Phys Med Rehabil. 2009 Dec;90(12):2019-25. doi: 10.1016/j.apmr.2009.08.139. PMID 19969163
- [Background] Toosizadeh N, Wahlert G, Fain M, Mohler J. The effect of vibratory stimulation on the timed-up-and-go mobility test: a pilot study for sensory-related fall risk assessment. Physiol Res. 2020 Aug 31;69(4):721-730. doi: 10.33549/physiolres.934451. Epub 2020 Jul 16. PMID 32672046
- [Background] Powden CJ, Hogan KK, Wikstrom EA, Hoch MC. The Effect of 2 Forms of Talocrural Joint Traction on Dorsiflexion Range of Motion and Postural Control in Those With Chronic Ankle Instability. J Sport Rehabil. 2017 May;26(3):239-244. doi: 10.1123/jsr.2015-0152. Epub 2016 Aug 24. PMID 27632835